CLINICAL TRIAL: NCT03897010
Title: Alveolar Ridge Augmentation Using Resorbable Bioactive Silica-calcium Phosphate Composite (SCPC): Clinical and Histology Evaluation
Brief Title: Evaluation of Silica-calcium Phosphate Composite in Socket Augmentation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Doaa Adel, Lecturer of Periodontology, Faculty of Dentistry, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 121812
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Ridge Deficiency
Keywords: Silica-calcium phosphate composite; Socket augmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Silica-calcium phosphate composite Group (Active Comparator): Participants underwent socket augmentation procedures and dental implant placement in a staged approach. Atraumatic extraction of badly decayed tooth was performed. The socket was debrided with curettes and alveolar spoons; the granulation tissue was carefully removed. Free gingival gingival graft (1.5 to 2 mm thick) was taken from the area between the first and second premolar, 5 mm from gingival margin. Bioactive porous SCPC dental bone graft granules in the size range 90-710 micron were mixed with saline and loosely packed in the extraction sockets as per the manufacturer. The grafted SCPC granules were covered with free gingival graft obtained from the palatal tissues and sutured to stabilize the grafting material in place.
  Interventions: Device: Socket Graft
- Control Group (Placebo Comparator): Participants underwent atraumatic extraction of badly decayed tooth was performed. The socket was debrided with curettes and alveolar spoons; the granulation tissue was carefully removed. The socket left to heal.
  Interventions: Device: Socket Graft

INTERVENTIONS:
Device: Socket Graft — 5 patients had bilateral decayed upper premolar or anterior teeth, in one side SCPC graft was inserted in socket and in the contralateral site was a control, 5 months months postoperative core biopsies were taken from both grafted sockets and control ungrafted sockets during implant insertion. The biopsy samples from SCPC-grafted and control ungrafted sockets were fixed, decalcified and embedded into paraffin wax. All samples were serially sectioned in serial 5μm-thin sections were stained separately with Hematoxylin and Eosin staining, Sirius red and Mason trichrome and immunostaining with osteopontin.
  Other Names: socket augmentation; Socket preservation

SUMMARY:
Ideal bone graft should possess osteogenic, osteoinductive, and osteoconductive properties. Unfortunately, all of these are solely found within the autogenous graft that is available only in limited quantities, and it is associated with substantial post-surgical morbidity, However in this study Silica-calcium phosphate composite (SCPC) confirmed clinically, radiographically, histomorphometricand immunohistochemically the vitality and functionality of the newly formed bone. Histology and immunohistochemistry demonstrated maturation of the newly formed bone as indicated by presence of osteocytes, Haversian systems, blood vessels, compact mineralized collagen type I and high immune staining for osteopontin.

DETAILED DESCRIPTION:
Alveolar ridge resorption following teeth extraction leads to 50% loss in bone width over one year period which corresponds to 5 -7 mm mainly from the buccal rather than palatal\lingual aspects. Several calcium phosphates from bovine and synthetics sources are used for preservation of extraction socket; however with variable degrees of success. The aim of the present study is to evaluate clinically, radiographically and histologically the effect of Silica-calcium phosphate composite (SCPC) granules on new bone formation qualitatively and quantitatively following socket augmentation. This case series study was performed in five (n = 5) participants (one male and four females), all participants underwent socket augmentation procedures and dental implant placement in a staged approach. All participants were fully informed about the procedures, including the surgery, bone substitute materials and implants. Each participant had one extraction socket to be grafted with silica-calcium phosphate SCPC dental bone graft granules and the contralateral socket served as ungrafted control. Clinical, radiographic and histological evaluation was assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients require extraction of bilateral non-restorable (premolar or anterior) tooth located in the maxillary arch and need implant restoration.
* Teeth to be extracted are free from acute periapical infection or active periodontitis.
* Buccal plate of bone is intact
* Systemic free patients
* Patients were able to swallow tablets.

Exclusion Criteria:

* Patients with remaining root accompanied with acute periapical infection or sinus tract
* Insulin dependent diabetes patients.
* Thyroid disease patients.
* Smoker´s patients
* Patients with compromised health (ASA (III or IV) - according to the classification of American Society of Anaesthesiology including drug or alcohol abuse or any significant systemic disease.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Clinical outcome | 5 months
  Clinical parameters on the tooth to be extracted in both test and control groups were assessed. Buccal gingival thickness was measured using clinical reference points 4 mm away from the gingival margin by a graduated periodontal probe.
Clinical outcome | 5 months
  Buccolingual bone width was measured by bone caliper 4 mm away from the gingival margins
Histological outcome | 7 months
  histomorphometric measurement of amount of residual graft percent and amount of new vital bone formation in the newly formed bone. The sections were obtained from the core biopsy in 5µm thickness and were stained by Hematoxylin and Eosin.

SECONDARY OUTCOMES:
Immunohistochemical analysis | 7 months
  Evaluation of Osteopontin expression in the newly formed bone.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adel-Khattab D, Afifi NS, Abu El Sadat SM, Aboul-Fotouh MN, Tarek K, Horowitz RA. Bone regeneration and graft material resorption in extraction sockets grafted with bioactive silica-calcium phosphate composite (SCPC) versus non-grafted sockets: clinical, radiographic, and histological findings. J Periodontal Implant Sci. 2020 Dec;50(6):418-434. doi: 10.5051/jpis.2000040002. PMID 33350181